CLINICAL TRIAL: NCT01996891
Title: Effects of an Anti-Inflammatory Diet on Pulmonary Function in Pediatric Asthma
Brief Title: Asthma (and Dietary) Inflammation Reduction
Acronym: AIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit adequate number of participants and high attrition rate
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, David S. Ludwig, MD, PhD, Director, Obesity Prevention Center, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 00006708
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: Asthma; Nutrition; Anti-inflammatory diet
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-Inflammatory Diet First (Other): For the first 6 weeks, subjects will receive the anti-inflammatory diet. For the second 6 weeks, subjects will consume their habitual diet.
  Interventions: Other: Anti-Inflammatory Diet
- Anti-Inflammatory Diet Second (Other): For the first 6 weeks, subjects will consume their habitual diet. For the second 6 weeks, subjects will receive the anti-inflammatory diet.
  Interventions: Other: Anti-Inflammatory Diet

INTERVENTIONS:
Other: Anti-Inflammatory Diet — The anti-inflammatory diet will focus on reducing glycemic load, and increasing fiber, fruits, vegetables, legumes and food-based omega-3 fatty acid content.

SUMMARY:
The purpose of this study is to evaluate the effects of a diet that is low in glycemic load and abundant in fiber, fruits, vegetables, legumes and omega-3 fatty acids ("anti-inflammatory diet") on pulmonary function in pediatric patients with asthma. The primary endpoint will be change in forced expiratory volume in one second in response to the diet intervention. Secondary outcomes will include additional spirometry measures, fraction of exhaled nitric oxide, and assessment of symptomatic asthma control. In addition, we will identify potential physiological mechanisms relating diet with lung function, including changes in systemic inflammation, insulin sensitivity, and intestinal microbiome composition.

DETAILED DESCRIPTION:
Asthma, an inflammatory disease of the airway mucosa, is highly correlated with obesity and nutritional intake in multiple cross-sectional studies. Limited interventional data in adults with asthma, relying on behavioral modification, have reported that asthma control significantly improves with caloric restriction and diets enriched with antioxidants, and may improve with increasing omega-3 fatty acid content. A comprehensive diet harnessing anti-inflammatory properties of multiple foods may have synergistic effects on bronchial inflammation and pulmonary function, yet this possibility remains largely untested, especially in children.

We propose a randomized, controlled cross-over trial, with 6-week treatment arms, in pediatric patients with moderate to severe asthma. The experimental diet will focus on reducing glycemic load, and increasing fiber, fruits, vegetables, legumes and food-based omega-3 fatty acid content. The comparison diet will be each participant's habitual diet. Both diets will be isocaloric and weight maintaining, to isolate the effects of the dietary composition from the known beneficial effects of weight loss. In addition, the home delivery of prepared meals will alleviate the variable and incomplete adherence commonly observed in behavioral studies.

ELIGIBILITY:
Inclusion Criteria:

* Age 10-21 years
* Clinical diagnosis of moderate or severe persistent asthma
* Currently prescribed inhaled corticosteroids for asthma with anticipated stable dosing regimen for the duration of the study
* Admission to Boston Children's Hospital for clinical asthma exacerbation
* Medical clearance from primary care provider
* Willingness to comply with study diet

Exclusion Criteria:

* Body mass index (BMI) < 3rd centile (age- and gender- adjusted normative range from Center for Disease Control)
* Known eating disorder
* Celiac disease
* Any food allergy
* Any other major illness as assessed by medical history or the following screening tests:
* Alanine aminotransferase (ALT) > twice upper limit of normal for age
* Creatinine > 1.0 mg/dL for age 10-18 years; > 1.2 mg/dL for females > 18 years; or > 1.4 mg/dL for males > 18 years)
* Random glucose > 200 mg/dL
* Hemoglobin < 11 g/dL for males age 10-18 years; < 11. g/dL for females age 10-18 years; <11.4 g/dL for males >18 years; or <10.9 g/dL for females age > 18 years
* Use of systemic steroids for indication other than asthma

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | End of 6-week intervention

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | End of 6-week intervention
Forced expiratory flow 25-75% (FEF25-75) | End of 6-week intervention
Fraction of exhaled nitric oxide (FeNO) | End of 6-week intervention
Asthma Control Questionnaire (ACQ) | End of 6-week intervention
Asthma Control Test (ACT) | End of 6-week intervention
Pediatric Asthma-Related Quality of Life Questionnaire | End of 6-week intervention
Asthma medication use | End of 6-week intervention
Serum inflammatory markers, including C-reactive protein (CRP), erythrocyte sedimentation rate (ESR), tissue necrosis factor-alpha (TNF-alpha), interleukin-6 (IL-6), plasminogen activator inhibitor-1 (PAI-1) | End of 6-week intervention
Asthma-related inflammatory markers, including eosinophilic cationic protein (ECP), monocyte chemoattractant protein (MCP-1) | End of 6-week intervention
Measures of insulin sensitivity, including fasting glucose, fasting insulin and adiponectin | End of 6-week intervention
Intestinal Microbiome Composition, including 16S sequencing and fecal short chain fatty acid levels | End of 6-week intervention
Serologic markers of nutritional status, including vitamin D | End of 6-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Bridget Hron, MD, Study Director — Boston Children's Hospital; Cara Ebbeling, PhD, Study Director — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States